CLINICAL TRIAL: NCT04858633
Title: Efficacy of Hydroxychloroquine (HCQ) as Post Exposure Prophylaxis (PEP) for Prevention of COVID-19 in Asymptomatic Individual at Risk for SARS-CoV-2 Infection-A Randomized Control Clinical Trial
Brief Title: Hydroxychloroquine (HCQ) as Post Exposure Prophylaxis (PEP) for Prevention of COVID-19
Acronym: PEP-CQ
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Deba Prasad Dhibar, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: INT/IEC/2021/SPL456
Record Dates: First submitted 2021-03-22; First posted 2021-04-26 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Covid19; COVID-19 Prevention
Keywords: Covid19, Hydroxychloroquine (HCQ)
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEP group (Active Comparator): Tablet HCQ 400 mg q 12 hourly on day one followed by 400 mg once weekly for 3 weeks (total 5 tablets, cumulative dose of 2000 mg)
  Interventions: Drug: Hydroxychloroquine (HCQ); Other: Standard care
- Control group (Placebo Comparator): Placebo one tablet 12 hourly on day one followed by one tablet once weekly for 3 weeks (total 5 tablets)
  Interventions: Other: Standard care; Other: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine (HCQ) — Tablet HCQ 400 mg q 12 hourly on day one followed by 400 mg once weekly for 3 weeks (total 5 tablets, cumulative dose of 2000 mg )
  Arms: PEP group
Other: Standard care — Standard therapy in the form of home quarantine for 2 weeks along with social distancing and personal hygiene
Other: Placebo — Tablet placebo one tablet 12 hourly on day one followed by one tablet once weekly for 3 weeks (total 5 tablets)
  Arms: Control group

SUMMARY:
COVID-19 affected more than 9 million of people with more than 130 thousand death in India. If adequate preventive and therapeutic measures are not taken, India has very high risk of affecting million of more people with high mortality because of the large population along with very high population density. At present there are no definitive therapeutic drugs or vaccine available for the treatment and prevention of SARS-CoV-2 infection. Symptomatic and supportive care are being given to COVID-19 cases along with isolation and quarantine measure are being taken for the suspected individual at risk for COVID-19 to limit the spread of the SARS-CoV-2 infection . Among the all the drugs being used for the treatment of COVID-19, hydroxychloroquine (HCQ), has given some rays of hope to battle against this deadly pandemic. HCQ has some anti viral effect against SARS-CoV in vitro. HCQ is quite safe and being used in rheumatology patients for lifelong without much side effect, so it allow for higher dose without any significant side effects and drug-drug interaction. Recently published clinical trial suggested HCQ can be used for the therapeutic purpose of the SARS-CoV-2 infection and many governments have endorsed that due to lack of any other better alternative drugs. Indian council of medical research (ICMR) has advised for HCQ prophylaxis for the people who are at risk for developing SARS-CoV-2 infection, all asymptomatic health care workers involved in taking care of suspected or confirmed COVID-19 cases and all asymptomatic household contacts of laboratory confirmed COVID-19 cases. With this encouragement an open level clinical trial was conducted on HCQ as post exposure prophylaxis (PEP) for the prevention of COVID-19 in asymptomatic high risk house hold contact of the laboratory confirmed COVID-19 cases. The result was very promising showing absolute risk reduction of around 9% in participant who received PEP with HCQ as compared to the control group and there was no serious adverse event. But there is still conflicting scientific data to prove or disprove the efficacy of HCQ for the treatment and prophylaxis for SARS-CoV-2 infection. Being a tertiary care center PGIMER is catering many states which include Punjab, hariyana, himachal Pradesh, Uttara khand, Uttar Pradesh. This put the institute to handle highest burden of suspected cases of SARS-CoV-2 in northern India. So, this double blind clinical trial has been planned to evaluate the efficacy of HCQ as PEP for the prevention of COVID-19 in asymptomatic individuals who are at risk for SARS-CoV-2 infection.

The asymptomatic individual with direct contact with laboratory confirmed COVID-19 cases will be randomized into one PEP group and one control/placebo group as per inclusion and exclusion criteria. Individual who will not give consent for HCQ prophylaxis and those with contraindication for HCQ therapy like, hypersensitivity to HCQ or 4-aminoquinolone derivatives, patients with known retionopathy, cardiac arrhythmia, G6PD deficiency, psoriasis and pregnancy will be excluded from the study. All symptomatic individual and all health care workers related to suspected or proven COVID-19 and who received CoVID-19 vaccine will be excluded from the study. The PEP group will receive tablet HCQ 400 mg q 12 hourly on day one followed by 400 mg once weekly for 3 weeks (total cumulative dose of 2000 mg). The control group will receive placebo instead of HCQ. Both the groups will receive standard care of therapy in the form of home quarantine for 2 weeks along with social distancing and personal hygiene. The participants will be followed up for 4 weeks telephonically or physically as and when required and will be enquired regarding development of any COVID-19 symptoms like fever, cough, sore throat, shortness of breath, diarrhoea, myalgia. During follow up nasopharyngeal swab of the participants will be taken for processing reverse transcription polymerase chain reaction (RTPCR) for the detection of SARS-CoV-2 RNA to confirm the CoVID-19. Samples for RTPCR will be taken when any asymptomatic participants becomes symptomatic and by the 5-14 days of contact in asymptomatic participants through in-hospital visit at the institute's COVID-19 screening clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Male/Female
2. Age of ≥18 years
3. Asymptomatic individual with direct contact with laboratory confirmed COVID-19 cases

Exclusion Criteria:

1. Symptomatic individual 2. Health care worker 3. Individual who will not give consent for HCQ prophylaxis 4. Contraindication for HCQ therapy 5. Pregnancy 6. Individual who received COVID-19 vaccine

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of COVID-19 | 4 weeks
  Both the definite and probable COVID-19 cases together are defined as COVID-19 case
Definite COVID-19 | 4 weeks
  Participant with RTPCR positive for SARS-CoV-2 and with or without symptoms will be defined as definite COVID-19 case
Probable COVID-19 | 4 weeks
  The participant with new onset symptoms, but RTPCR negative for SARS-CoV-2 or cannot be performed for any reason will be defined as probable COVID-19 case.

SECONDARY OUTCOMES:
New onset symptoms of COVID-19 | 4 weeks
  Incidence of new onset symptoms of COVID-19 in asymptomatic participants
Compliance | 4 weeks
  Percentage of participants will be completing the advised therapy
Adverse drug reaction (ADR) | 4 weeks
  Incidence of adverse drug reaction among the participants

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No
All data requests should be submitted to the PI (DPD) for consideration. Data sharing may be considered by the PI after due approval from IEC.